CLINICAL TRIAL: NCT06292910
Title: Predictability of Central Venous to Arterial CO2 Difference (AVCO2) in Children With Cardiac Surgery to Poor Outcomes
Brief Title: Central Venous to Arterial CO2 Difference and Low Cardiac Output Syndrome Related Outcomes in Children After Cardiac Surgery
Acronym: VACO2
Status: Completed | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Pharsai Prasertsan, Assist. Prof, Prince of Songkla University
Other Study IDs: REC 64-299-1-1
Record Dates: First submitted 2024-02-09; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Congenital Heart Disease; Perioperative/Postoperative Complications; Lactate Blood Increase
MeSH Terms: conditions — Heart Defects, Congenital; Postoperative Complications; Hyperlactatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: arterial and central venous blood gas analysis, lactate — blood gas analysis

SUMMARY:
The goal of this clinical trial is to compare the capability of 3 different bedside surrogates in children who underwent cardiac surgery and were admitted in intensive care unit. These test are lactate, oxygen saturation from central venous and the carbon dioxide gap between central venous and arterial.

The main questions is which one is the best prognostication for post operation poor outcomes Participants will be taken routine blood test for post cardiac care (at ICU arrival, 6, 12, and 24 hour post operation) and follow the their outcomes. There is no any intervention or drug in this research

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-18 years old with either congenital or acquired cardiac disease
* Undergone cardiopulmonary bypass for cardiac surgery
* Be admitted in PICU for post-operative care

Exclusion Criteria:

* Preterm infant (GA < 37 weeks) or weight less than 2 kg
* Patient who weaned off cardiopulmoanry bypass and required extracorporeal membrane oxygenator (ECMO) before leaving the operating room
* Patient who required emergency cardiac operation within 24 hour after hospitalization
* Patient who had significant residual left side outflow tract obstruction (e.g., coarctation of aorta, interrupted aortic arch) which defined by difference of SBP between upper and lower extremities more than 10 mmHg
* Patient who had already participated in another research project
* Patient who does not have both arterial line and central line catheter back from operating room
* Parents or legal guardian refuse to inform consent.

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with cardiac disease in Songklanagarind hospital who undergone open cardiac surgery with cardiopulmonary bypass (age < 18 years old)
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2021-08-08 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
number of participant who developed low cardiac output syndrome related poor outcomes within 24 hour post operation | from time of subject was admitted to ICU until the 24 hour post operation
  the low cardiac output syndrome (LCOS) related poor outcomes was diagnosed if at least two of the following criteria were met within 24 hours postoperatively:
  1. clinical LCOS: prolonged capillary refill >3 seconds, systolic blood pressure <5th percentile for age and sex, persistent elevation of left atrial pressure >10 mmHg for at least 6 hours, and low urinary output (<1 mL/kg/hour) for at least 6 hours despite diuretic use
  2. laboratory LCOS: persistently elevated lactate level (>2 mmol/L), metabolic acidosis with an increase in the base deficit (>4 mmol/L) for at least 6 hours consecutively
  3. Vasoactive-inotropic score ≥20
  4. any unplanned surgery or intervention, cardiac arrest, or utilization of ECMO
  5. left ventricular fraction <50% on echocardiography

SECONDARY OUTCOMES:
ventilator days | from date of subject was admitted to ICU until the date of subject was extubated, assessed up to 28 days
  number of the days subject was intubated and used mechanical ventilator after operation
inotrope days | from date of subject was admitted to ICU until the date of subject was free of inotropic drugs, assessed up to 28 days
  number of the days subject was on inotropic medication after operation
length of stay in ICU | from date of subject was admitted to ICU until the date of subject was discharge, assessed up to 28 days
  number of the days subject was stay in ICU after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
This data might be analyzed in other project and also we need to submit the form of data sharing to local EC unit.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT06292910/Prot_SAP_000.pdf